CLINICAL TRIAL: NCT01785511
Title: Does Ultraviolet Irradiation Reduce Platelet Reactivity and Improve Coronary Microvascular Function in Man?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UVA Study
Record Dates: First submitted 2012-06-20; First posted 2013-02-07 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Hypertension
Keywords: hypertension; UV radiation; coronary flow reserve; nitric oxide
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham UVA (Sham Comparator): sham exposure will be provided by covering the UVA lamps with space blanket.
  Interventions: Radiation: UVA Radiation
- UVA Radiation (Experimental): Patients will be exposed to UVA radiation for 20 minutes
  Interventions: Radiation: UVA Radiation

INTERVENTIONS:
Radiation: UVA Radiation — UVA radiation exposure for 20 minutes

SUMMARY:
Endothelium derived nitric oxide (NO) regulates vascular tone and blood pressure in man. NO also inhibits platelet aggregation and mediates a variety of beneficial anti-inflammatory and repair mechanisms. NO may also be a mediator in the release of the endogenous fibrinolytic factor, tissue-plasminogen activating factor (t-PA) from the endothelium.1 Via these actions it plays a very important role in protection of the vasculature from atherothrombosis and clinical sequelae such as myocardial infarction and stroke.

Visible and ultraviolet (UV) light relax vascular smooth muscles by producing NO in a phenomenon known as photorelaxation.2 The investigators have demonstrated significant stores of pre-formed, bound NO and other nitrosospecies in human skin, which are rapidly released upon exposure to UVA.3 The investigators have demonstrated recently that serum nitrite and nitroso-species are increased after standing in a UVA phototherapy cabinet and that local UVA exposure is associated with increased forearm arterial blood flow that is independent of skin temperature. The investigators have also demonstrated a fall in mean arterial blood pressure in subjects exposed UVA.

Cardiovascular morbidity and the prevalence of hypertension vary with latitude. The investigators hypothesise that some of this geographical variation may be explained by a diminished sunlight/UVA exposure with attendant negative effects upon NO bio-availability.4 To further examine the potential beneficial effects of UVA exposure we will examine the effects of whole-body UVA upon platelet activation and upon myocardial/coronary arterial flow reserve. The investigators will correlate these measures with systemic nitrate, nitrite and nitroso-species content in healthy volunteers.

HYPOTHESES

1. UVA irradiation enhances coronary flow reserve in healthy volunteers.
2. UVA irradiation suppresses platelet activation in healthy volunteers.
3. UVA irradiation enhances the release of endogenous fibrinolytic factors in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged between 18-45 years (inclusive).

Exclusion Criteria:

* Inability to provide informed consent
* Co-existent systemic disease (including any history of asthma, reactive airways disease or hypertension)
* Contraindication to UVA treatment
* Any history of cardiac conduction abnormality (including bundle branch block or atrial fibrillation)
* Smoker
* Current intake of aspirin, other non-steroid anti-inflammatory medications or any regular medication.
* Recent infective/inflammatory condition
* Echocardiographic evidence of left ventricular hypertrophy (left ventricular septal diameter >1.2 cm in diastole), systolic dysfunction or significant valvular stenosis or regurgitation.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Coronary Flow Reserve | 0, 20, 40 and 60 mins
  Change in coronary flow assessed pre and post UVA radiation versus control

SECONDARY OUTCOMES:
Platelet Activation | 0, 20, 40 and 60 mins
  Platelet activation assessed using platelet monocyte activity
Endogenous Fibrinolysis | 0, 20, 40 and 60 minutes
  Assessed using flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Ninian Lang, MbChB, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Lothian, United Kingdom